CLINICAL TRIAL: NCT06927323
Title: Effects of Otago Exercise Program Combined With Action Observation Training on Balance, Gait and Functional Activities in Post Stroke Patients
Brief Title: Otago Exercise Program Combined With Action Observation Training in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0243 Rimsha Ashfaq
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Action observation training, Otago exercises, Stroke, Gait, Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A. Otago Exercise Program (Experimental): The Otago Exercise Program (Group A) includes specific exercises for strength and balance improvement. These exercises were conducted three times a week. Each training session lasted for 35-40 minutes.
  Interventions: Other: Otago exercise program
- B. Action Observation Training combined with Otago exercise program (Experimental): Participants will be instructed to watch a video on a 22-inch screen positioned 1 meter away from them, while comfortably seated in a chair with armrests. They are not allowed to follow along or engage in any movement while watching the video. The duration of the video viewing will be 17 minutes (1 minute for each video), followed by a 35-minutes of exercise (2 minutes maximum per session).
  Interventions: Other: Otago exercise program

INTERVENTIONS:
Other: Otago exercise program — The Otago Exercise Program is composed of strength training and balance training. Strength training consisted of flexion and extension exercises of the knee, ankle, and toe joints, as well as hip opening exercises to strengthen the sides of the pelvis. Balance training consisted of walking backwards, walking in a figure of eight, heel-toe walking, standing on one leg, walking on the heels, walking on the toes, heel-toe walking backwards, standing up from a sitting position, and walking up stairs. Otago exercise program will be performed with action observation train will be instructed to watch a video on a 22-inch screen positioned 1 meter away from them, while comfortably seated in a chair with armrests. They are not allowed to follow along or engage in any movement while watching the video.
  Other Names: Action Observation Training combined with Otago exercise program

SUMMARY:
Stroke is one of the main causes of adult disability worldwide and global health problem. Due to ongoing neurological sequelae post stroke patients have a two-fold higher risk of falling than other people with same age or gender. As the stroke patients, balance is impaired and can lead to complications such as fall. Promising interventions that could be beneficial to improve the aspects of gait and balance include Otago exercises and Action observation training. The objective of this study is to determine the effects of Otago exercise combined with Action observation (AO) training on the balance, gait and functional activities in post stroke patients.

A double-blinded randomized control trial will be conducted at Rehabilitation centers, outpatient clinics, and Hospitals for ten months. The sample size will consist of 60 participants. Participants which meet the inclusion criteria will be taken through non-probability convenience sampling technique. Participants will be randomly assigned into two groups: 30 to action observation (AO) training plus Otago exercise group (n= 30) and 30 to Otago exercise group (n= 30). The AO plus Otago and Otago groups will be performed 35 to 40 minutes of strength training and balance exercises from the Otago Exercise Program 3 times a week for 12 weeks. Data will be collected through various assessment tools including Berg Balance Scale (for balance), Dynamic gait index (for gait) and Functional Independence Measure (for functional activities). The effects of the interventions will be measured at pre-treatment and post-intervention. Paired t-test will be adopted to find the statistical difference within the groups and independent t-test will be applied to find the statistical difference between the groups. Data analysis will be performed by using SPSS 26 software.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling given criteria will be included in this study

* Both male and female participants will be included
* The age limit for the participants will be 40-65 years
* Sub-acute and chronic ischemic stroke up to 2 years.
* Participants with BBS score between 35-40.
* Participants having Montreal Cognitive Assessment (MoCA) score greater than 24 (out of 30).
* Participants can walk with or without assistance.

Exclusion Criteria:

Participants having given criteria will be excluded from this study

* Participants with other neurological diseases.
* Participants who will not be able to understand the informed consent form.
* Participants already involved in an exercise program for fall prevention.
* Participants have no visual field defect, no abnormality in the vestibular organs, no orthopedic disease, and an unrestricted range of motion.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (for balance) | 8 weeks
  The BBS is constructed to assess balance ability of older people and identify their risk for falling. The BBS is a 14-task scale that requires subjects to maintain their balance in positions and tasks of increasing difficulty. Specific components of the BBS parallel some gait requirements such as unsupported leg stance and standing with 1 foot in front of the other. Other components address tasks such as rising to stand or standing unsupported. It has an ordinal scale of 0 to 4 points (best performance, 56). The BBS is well documented and has strong psychometric properties for people with stroke. For subjects with stroke, the interrater and intrarater reliability were found to be .97 and .98, respectively. A score of 44 or less has been found to indicate a higher risk of falls.
Dynamic Gait Index (for gait) | 8 weeks
  The DGI is 8 items test that includes walking, walking while changing speed, walking while turning the head horizontally and vertically, walking with pivot turn, walking over and around obstacles, and stair climbing. The scoring of the DGI is based on a 4-point scale ranging from 0 to 3, with 0 indicating severe impairment and 3 indicating normal ability. The best performance total score is 24. A low composite DGI score thus indicates greater impairment in functional mobility. The DGI has been found to be reliable and valid for older people (.96) (ICC.98). Scores of or below 19 points on the DGI indicate a risk of falling in older people and a score of less than 12 points discriminated between fallers and non-fallers.
Functional Independence Measure (for functional activities) | 8 weeks
  The FIM instrument is a minimum data set that measures 18 functional activities, 13 of which involve motor activities and 5 of which involve cognitive activities. The tool has a 7-level scale for scoring each of the items. For example, a score of 1 means that a patient is dependent and is able to provide less than 25% of the effort for a given activity, and a score of 7 means that a patient is completely independent and can perform an activity without assistive devices in a safe and timely manner.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No